CLINICAL TRIAL: NCT05906589
Title: Exploring Mechanism of Action of Dietary Fibre on the Gut Microbiota and Metabolites: Can we Identify Responders and Non-responders to Psyllium and Inulin Dietary Fibres?
Brief Title: Exploring Mechanism of Action of Dietary Fibre on the Gut Microbiota and Metabolites
Acronym: MERLIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 501
Record Dates: First submitted 2023-05-19; First posted 2023-06-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Psyllium; Inulin
Keywords: Dietary fibre; Dietary fiber; Gut microbiota
MeSH Terms: interventions — Inulin; Psyllium; ispaghula seed; maltodextrin

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to one of the 6 different intervention combinations for the supplements ((A) placebo; (B) inulin; (C) psyllium plus inulin) with the same number of participants in each of the combinations.
  There are 6 possible combinations:
  * A > B > C
  * B > A > C
  * C > B > A
  * A > C > B
  * C > A > B
  * B > C > A
Who Masked: Participant, Investigator
Masking Description: The study will be double blind, meaning both the investigator and the participants will not know if the participants are receiving inulin, psyllium plus inulin or the placebo. However, there is some difference in the consistency of the powders. The supplements will be labelled A, B and C by an independent party otherwise not involved in the study, and the investigator and participants will not know which supplement is which letter during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inulin (Experimental): The participant will be asked to administer the provided doses of 8g inulin twice daily.
  Interventions: Dietary Supplement: Inulin
- Inulin + psyllium (Experimental): The participant will be asked to administer the provided doses of 8g inulin + 3.5g psyllium twice daily.
  Interventions: Dietary Supplement: Inulin; Dietary Supplement: Psyllium
- Maltodextrin (Placebo Comparator): The participant will be asked to administer the provided doses of 8g maltodextrin twice daily.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Inulin — The participant will take inulin twice daily over a 14 day period.
  Arms: Inulin; Inulin + psyllium
Dietary Supplement: Psyllium — The participant will take psyllium twice daily over a 14 day period.
  Other Names: Ispaghula husk
  Arms: Inulin + psyllium
Dietary Supplement: Maltodextrin — The participant will take maltodextrin twice daily over a 14 day period.
  Arms: Maltodextrin

SUMMARY:
Cancer patients receiving pelvic radiotherapy suffer side effects to the intestine, including diarrhoea and occasionally rectal bleeding, often worsened by chemoradiation. Many pelvic radiotherapy patients receive a form of dietary fibre, psyllium husk, to manage their diarrhoeal symptoms. There is evidence in mice that dietary fibre supplementation can improve tumour response and reduce normal tissue side effects caused by radiation. If this were to be confirmed in humans, it would be a major advance in patient treatment. The investigators will conduct a study in healthy subjects to assess mechanisms and response to dietary fibre.

The investigators will conduct a within-subject diet intervention study on healthy older adults (>60 years old) to determine if a subset of the population are responders to dietary fibre manipulation, using inulin with or without psyllium. This will allow assessment of the physiological impact of dietary fibre. Participants will receive placebo, inulin, or psyllium plus inulin in random order (6 possible combinations) for two weeks each with two-week washout periods.

Baseline faecal microbial activity, short chain fatty acid (SCFA) concentrations, and habitual fibre intake, determined by dietary questionnaires/food diaries will be used to identify individuals in whom dietary fibre manipulation might have a positive impact. Individuals who respond to dietary fibre supplementation may be found to have elevated levels of some SCFAs and significantly increased relative abundance of certain microbiota. Dietary parameters, bacterial relative abundance and SCFA levels will be correlated with plasma cytokine levels.

DETAILED DESCRIPTION:
Of all patients receiving radiotherapy for cancer in 2018 and 2019, 28.6% were treated for a pelvic malignancy. The dose of radiotherapy necessary to cure the tumour often causes side effects in the surrounding healthy tissues, which can significantly impact the patients quality of life. Chemoradiation, the addition of chemotherapy to radiotherapy, improves tumour cure rates by radiosensitising the tumour, but at the expense of worsened normal tissue effects. Most patients over 80 years are unable to tolerate chemoradiation. With an aging population, there is an urgent clinical need to find alternatives to chemoradiation.

A difference in the composition and diversity of the gut microbiota has been found in responders versus non-responders to immunotherapy and in patients experiencing different levels of toxicities following radiotherapy. This indicates that the microbiota could be used to predict, prevent, or treat radiation enteropathy. An often-found side effect in pelvic radiotherapy patients is diarrhoea. Many pelvic radiotherapy patients receive a form of dietary fibre, known as psyllium husk (ispaghula husk or FybogelTM) to manage their diarrhoeal symptoms. Dietary fibres like psyllium and inulin are non-digestible carbohydrates found in fruits, vegetables, whole grains and legumes. They are anaerobically fermented by the gut bacteria, producing SCFAs, including acetate, propionate, and butyrate. SCFAs are the main performers in the interplay between diet, microbiota and health, and have anti-inflammatory and also anti-tumorigenic properties.

A high intake of dietary fibre is proven to decrease the risk of type 2 diabetes, colon cancer and cardiovascular disease by reducing the digestion and absorption of macronutrients and decreasing the contact time of carcinogens with the intestinal lumen. There is emerging evidence that the inclusion of dietary fibre supplements in the diet could modify the tumour response to radiotherapy. If confirmed in humans, this would be a major advance in patient treatment.

In a mouse model of colitis, exhibiting similar acute symptoms to those due to radiotherapy, the addition of psyllium in the diet reduced colonic inflammation and protected intestinal tight junctions. This prevented penetration of luminal inflammatory molecules through the gut wall. In a similar model system, psyllium reduced the severity of colitis in C57BL/6 specific pathogen-free and germ-free mice, via microbiota-dependent and independent mechanisms.

Inulin, another dietary fibre, is rapidly fermented in the proximal large intestine. Here, it selectively increases the growth of the butyrate producer Faecalibacterium prausnitzii and Bifidobacterium spp.. Bifidobacteria are associated with anti-tumour effects and augmented dendritic cell function leading to increased Cytotoxic T-cell (CD8+) priming and accumulation in the tumour microenvironment.

The investigators found promising preliminary data in our mouse studies, indicating that psyllium with inulin enhances tumour control. Immunodeficient mice fed a 10% inulin diet had an improved tumour control following 6 gray (Gy) ionising radiation. Immunocompetent mice showed a delayed tumour growth when receiving psyllium plus inulin when compared to a normal or low fibre diet, accompanied by significantly increased tumour infiltration of cytotoxic T cells. Psyllium plus inulin also significantly increased the percentage of intestinal remaining after 14 Gy compared to a low fibre diet or psyllium alone. A psyllium plus inulin diet also modified intestinal immunity, particularly B cells. Furthermore, in mouse bladder cancer cell UPPL 1591-derived allografts, CD8+ (cytotoxic) T cells scored higher for psyllium and psyllium plus inulin than psyllium plus resistant starch. However, compared to humans, inbred mice are genetically more similar and are held in controlled environmental conditions, so humans are likely to demonstrate more variability in response to dietary fibre intervention.

The investigators will study a group of human participants to assess tolerance and responses to inulin and psyllium plus inulin, in terms of intestinal side effects, significant alterations in the microbiota, levels of SCFAs in plasma and faeces, and plasma inflammatory cytokines. The investigators will also investigate whether responders and non-responders within the study can be identified from baseline dietary information and/or microbial activity (based on faecal SCFA measurements), as an individual's current diet will influence their response to dietary fibre modification.

ELIGIBILITY:
Inclusion Criteria:

* >60 years old

Exclusion Criteria:

Medication exclusion criteria:

* Oral antibiotic use (within the past 3 months due to impact on gut microbiota).
* Anti-coagulants (Warfarin).
* Carbamazepine (epilepsy)
* Digoxin (heart conditions)
* Mesalazine (gut problems)
* Regular use of anti-constipation medication/laxatives.

Medical exclusion criteria:

* Food allergies, self-reported food sensitivity or intolerance.
* Type 1 or Type 2 diabetes.
* Coeliac disease or gluten intolerance.
* Metformin intake.
* Bowel obstruction
* Muscle weakness of the bowel
* Phenylketonuria.

Other exclusion criteria:

* Anyone with unsuitable veins for blood sampling.
* Anyone with chronic constipation (>3 days without defaecation).
* Anyone who is unable to fluently speak, read and understand English.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Microbial composition using 16S sequencing | 11 weeks per participant
  To explore the effect of inulin and psyllium plus inulin on microbial composition at baseline and after a 14-day intervention.
Short Chain Fatty Acid (SCFA) levels | 11 weeks per participant
  To explore the effect of inulin and psyllium plus inulin on short chain fatty acid levels at baseline and after a 14-day intervention.

SECONDARY OUTCOMES:
Tolerability of Inulin defined by questionnaire 'quality of life' and 'gastrointestinal wellbeing' | 11 weeks per participant
  To determine if 16 g inulin with or without 7 g psyllium dietary interventions are tolerable in older adults (>60 years old) assessed by completing gastrointestinal wellbeing questionnaires and quality of life questionnaires (SF36).
Tolerability of psyllium defined by questionnaire 'quality of life SF36' and 'gastrointestinal wellbeing' | 11 weeks per participant
  To determine if 16 g inulin with or without 7 g psyllium dietary interventions are tolerable in older adults (>60 years old) assessed by completing gastrointestinal wellbeing questionnaires and quality of life questionnaires (SF36).
Rate of habitual fibre intake before and during the intervention | 11 weeks per participant
  To determine if Food Frequency Questionnaires/3- day weighed food diaries (to assess habitual fibre intake before and during the intervention) can identify individuals in whom dietary fibre supplementation would have a positive impact on microbiota composition and SCFA levels.
Faecal SCFA concentrations | 11 weeks per participant
  Identify individuals in whom dietary fibre supplementation would have a positive impact using baseline faecal microbial activity (determined by faecal SCFA concentrations).
Elevated plasma SCFAs | 11 weeks per participant
  Change in SCFA levels in plasma from baseline in individuals that respond to dietary fibre supplementation after 14 days.
A 0.5 log10 change in health-associated Bifidobacterium spp. from baseline | 11 weeks per participant
  Detecting a 0.5 log10 change in health-associated Bifidobacterium spp. from baseline in individuals given psyllium plus inulin using faecal quantitative polymerase chain reaction.
Plasma cytokine IL-6 | 11 weeks per participant
  To determine if dietary parameters, bacterial relative abundances and SCFA levels are correlated with plasma cytokine IL-6 level (cytokine level will only be measured at the end of each intervention), which may influence radiotherapy outcomes in terms of tumour response and normal tissue effects.
Plasma cytokine IL-8 | 11 weeks per participant
  To determine if dietary parameters, bacterial relative abundances and SCFA levels are correlated with plasma cytokine IL-8 level (cytokine level will only be measured at the end of each intervention), which may influence radiotherapy outcomes in terms of tumour response and normal tissue effects.
Immunoglobulin A (IgA) and calprotectin levels | 11 weeks per participant
  To determine if the interventions alter gut health and inflammation, measured by faecal IgA and calprotectin at the end of each of the three interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Kiltie, Prof, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No.

REFERENCES:
- [Background] Wang L, Wang X, Zhang G, Ma Y, Zhang Q, Li Z, Ran J, Hou X, Geng Y, Yang Z, Feng S, Li C, Zhao X. The impact of pelvic radiotherapy on the gut microbiome and its role in radiation-induced diarrhoea: a systematic review. Radiat Oncol. 2021 Sep 25;16(1):187. doi: 10.1186/s13014-021-01899-y. PMID 34563216
- [Background] Bishehsari F, Engen PA, Preite NZ, Tuncil YE, Naqib A, Shaikh M, Rossi M, Wilber S, Green SJ, Hamaker BR, Khazaie K, Voigt RM, Forsyth CB, Keshavarzian A. Dietary Fiber Treatment Corrects the Composition of Gut Microbiota, Promotes SCFA Production, and Suppresses Colon Carcinogenesis. Genes (Basel). 2018 Feb 16;9(2):102. doi: 10.3390/genes9020102. PMID 29462896
- [Background] Carretta MD, Quiroga J, Lopez R, Hidalgo MA, Burgos RA. Participation of Short-Chain Fatty Acids and Their Receptors in Gut Inflammation and Colon Cancer. Front Physiol. 2021 Apr 8;12:662739. doi: 10.3389/fphys.2021.662739. eCollection 2021. PMID 33897470
- [Background] Tan J, McKenzie C, Potamitis M, Thorburn AN, Mackay CR, Macia L. The role of short-chain fatty acids in health and disease. Adv Immunol. 2014;121:91-119. doi: 10.1016/B978-0-12-800100-4.00003-9. PMID 24388214
- [Background] Kaczmarczyk MM, Miller MJ, Freund GG. The health benefits of dietary fiber: beyond the usual suspects of type 2 diabetes mellitus, cardiovascular disease and colon cancer. Metabolism. 2012 Aug;61(8):1058-66. doi: 10.1016/j.metabol.2012.01.017. Epub 2012 Mar 7. PMID 22401879
- [Result] Olopade FA, Norman A, Blake P, Dearnaley DP, Harrington KJ, Khoo V, Tait D, Hackett C, Andreyev HJ. A modified Inflammatory Bowel Disease questionnaire and the Vaizey Incontinence questionnaire are simple ways to identify patients with significant gastrointestinal symptoms after pelvic radiotherapy. Br J Cancer. 2005 May 9;92(9):1663-70. doi: 10.1038/sj.bjc.6602552. PMID 15856043
- [Result] Gopalakrishnan V, Helmink BA, Spencer CN, Reuben A, Wargo JA. The Influence of the Gut Microbiome on Cancer, Immunity, and Cancer Immunotherapy. Cancer Cell. 2018 Apr 9;33(4):570-580. doi: 10.1016/j.ccell.2018.03.015. PMID 29634945
- [Result] Reis Ferreira M, Andreyev HJN, Mohammed K, Truelove L, Gowan SM, Li J, Gulliford SL, Marchesi JR, Dearnaley DP. Microbiota- and Radiotherapy-Induced Gastrointestinal Side-Effects (MARS) Study: A Large Pilot Study of the Microbiome in Acute and Late-Radiation Enteropathy. Clin Cancer Res. 2019 Nov 1;25(21):6487-6500. doi: 10.1158/1078-0432.CCR-19-0960. Epub 2019 Jul 25. PMID 31345839
- [Result] Ogata M, Ogita T, Tari H, Arakawa T, Suzuki T. Supplemental psyllium fibre regulates the intestinal barrier and inflammation in normal and colitic mice. Br J Nutr. 2017 Nov;118(9):661-672. doi: 10.1017/S0007114517002586. PMID 29185927
- [Result] Llewellyn SR, Britton GJ, Contijoch EJ, Vennaro OH, Mortha A, Colombel JF, Grinspan A, Clemente JC, Merad M, Faith JJ. Interactions Between Diet and the Intestinal Microbiota Alter Intestinal Permeability and Colitis Severity in Mice. Gastroenterology. 2018 Mar;154(4):1037-1046.e2. doi: 10.1053/j.gastro.2017.11.030. Epub 2017 Nov 23. PMID 29174952
- [Result] Ramirez-Farias C, Slezak K, Fuller Z, Duncan A, Holtrop G, Louis P. Effect of inulin on the human gut microbiota: stimulation of Bifidobacterium adolescentis and Faecalibacterium prausnitzii. Br J Nutr. 2009 Feb;101(4):541-50. doi: 10.1017/S0007114508019880. Epub 2008 Jul 1. PMID 18590586
- [Result] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Result] Then CK, Paillas S, Wang X, Hampson A, Kiltie AE. Association of Bacteroides acidifaciens relative abundance with high-fibre diet-associated radiosensitisation. BMC Biol. 2020 Aug 19;18(1):102. doi: 10.1186/s12915-020-00836-x. PMID 32811478
- [Result] Walker AW, Ince J, Duncan SH, Webster LM, Holtrop G, Ze X, Brown D, Stares MD, Scott P, Bergerat A, Louis P, McIntosh F, Johnstone AM, Lobley GE, Parkhill J, Flint HJ. Dominant and diet-responsive groups of bacteria within the human colonic microbiota. ISME J. 2011 Feb;5(2):220-30. doi: 10.1038/ismej.2010.118. Epub 2010 Aug 5. PMID 20686513